CLINICAL TRIAL: NCT04722159
Title: Clinical Outcome of Patients With Resistant Hypertension Undergoing Renal Denervation: A Report From the Swedish Registry for Renal Denervation
Brief Title: Clinical Outcome of Patients With Resistant Hypertension Undergoing Renal Denervation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: ERP-2018-11640
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Hypertension, Renal
MeSH Terms: conditions — Hypertension, Renal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Treatment resistent hypertensives, treated with renal denervation: Patients having undergone renal denervation and fulfilling the criteria for resistant hypertension according to the criteria as applied in the Swedish Registry for Renal Denervation (Office BP >140/90 despite treatment with at least three antihypertensive drugs) with a follow up period of at least 5 years.
  Interventions: Device: Renal denervation
- Treatment resistent hypertensives, conservatively treated: Patients fulfilling the criteria for resistant hypertension according to the criteria as applied in the Swedish Registry for Renal Denervation (Office BP >140/90 despite treatment with at least three antihypertensive drugs) with a follow up period of at least 5 years.

INTERVENTIONS:
Device: Renal denervation — Catheter-based inhibition of renal sympathetic nerve traffic.
  Groups: Treatment resistent hypertensives, treated with renal denervation

SUMMARY:
Studies on the impact of RDN on cardiovascular surrogate markers have shown a variety of beneficial effects: RDN is associated with a decrease blood pressure (BP), left ventricular mass (LVM), a reduction in aortic pulse-wave velocity and BP variability as well as an increase in heart rate-recovery. Several of these aspects have been observed independently of office BP response, and might be mediated by a direct modulation of the sympathetic nervous system. Moreover, several independent real - world registries have shown an association of renal denervation and sustained blood pressure reductions of clinically relevant magnitude up to 36 months of follow - up.

Whether the sum of these effects may translate into an improvement of clinical outcomes remains unclear and constitutes the primary subject of proposed registry based study.

DETAILED DESCRIPTION:
Two registries interlinked by the Swedish personal identification number The Swedish Registry for Renal Denervation: The Swedish Registry for Renal Denervation is an investigator - initiated academic online database, developed by our group and supported by the Swedish authorities. The registry contains 130 variables summarizing baseline patient characteristics, procedural details, as well as follow - up data. The database contains patient data from the seven Swedish university hospitals that have performed RDN since 2011 exclusively, thereby providing a nation-wide data set with a follow-up of up to five years.

The Swedish Primary Care Cardiovascular Database (SPCCD):

SPCCD comprises data from 75 000 patients diagnosed with hypertension collected at primary care centres in the Stockholm and Skaraborg region during the time period 2001-2008. Patient baseline characteristics may be derived from the individual electronic medical records.

Study objectives:

* To describe the incidence of the composite end-point of myocardial infarction, stroke, heart failure and cardiovascular death in patients with resistant hypertension treated with RDN as compared to conservatively treated resistant hypertensives.
* Our hypothesis is that RDN treated individuals will show a lower event rate in regard to the composite clinical end - point during the first 5 years of follow - up when compared to conservatively treated individuals with resistant hypertension.

Inclusion criteria:

- Patients fulfilling the criteria for resistant hypertension according to the criteria as applied in the Swedish Registry for Renal Denervation (Office BP >140/90 despite treatment with at least three antihypertensive drugs) with a follow up period period of at least 5 years (SPCCD).

Methods and statistical analysis:

The primary end point of this study is the composite of myocardial infarction, stroke, heart failure and cardiovascular death in patients with resistant hypertension having undergone renal denervation (n = 300), compared to a control group of conservatively treated resistant hypertensives from the SPCCD. The necessary information about the diagnose codes for the events relevant for the primary end - point is made possible through the unique Swedish personal identification number and available through the Swedish population based registries for both the case - and control - group.

In order to adjust for differences in the baseline variables age, sex, diabetes, coronary artery disease, heart failure, baseline blood pressure, duration of hypertension, number of hypertensive drugs, we will perform a propensity score matched analysis which will be performed in 1 : 3 fashion.

Potential significance Despite the promising results of RDN in regard to several clinically relevant surrogate markers, including blood pressure, there are no outcome data available in the literature. Thus, the findings of this study may provide novel insights into the clinical effects of renal denervation and assess whether the sum of the previously observed beneficial effects may translate into an improved clinical outcome.

ELIGIBILITY:
Inclusion criteria:

Patients registered in the Swedish Registry for Renal Denervation or SPCCD, fulfilling the criteria for resistant hypertension according to the criteria as applied in the Swedish Registry for Renal Denervation (Office BP >140/90 despite treatment with at least three antihypertensive drugs).

Exclusion criteria:

Any patient who has withdrawn consent from being in either registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with resistant hypertension, registered in either the The Swedish Registry for Renal Denervation or the Swedish Primary Care Cardiovascular Database (SPCCD).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of the composite end-point of myocardial infarction, stroke, heart failure and death | From inclusion into the registry and 6 years forward
  Incidence of the composite end-point of myocardial infarction, stroke, heart failure and death

CONTACTS AND LOCATIONS:
Overall Officials: Bert Andersson, Study Chair — Sahlgrenska University Hospital
Locations (1):
- Sahlrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided